CLINICAL TRIAL: NCT03986060
Title: Shouldice Hospital Outcome Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: York University (Other)
Responsible Party: Principal Investigator, Joel Katz, Professor, York University
Other Study IDs: 1
Record Dates: First submitted 2019-06-12; First posted 2019-06-14 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective cohort study recruiting participants from the Shouldice Hospital. The study population consists of healthy patients electing to receive hernia surgery for a primary inguinal hernia on an inpatient basis. The goal of this study is to determine the incidence of hernia pain and its intensity as well as other related outcomes up to one year after primary unilateral inguinal hernia repair.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form.
* Willing to comply with all study procedures and be available for the duration of the study (patients have fixed address, access to phone, email, internet, and/or a computer)
* Male or female, aged 18 to 90 years.
* Subjects having surgery on a primary unilateral inguinal hernia
* In good general health as evidenced by medical history
* Capable of speaking and reading English sufficiently well to complete the questionnaires

Exclusion Criteria:

* Surgery is deemed an emergency procedure (any obstruction, incarceration or irreducible hernias).
* Other abdominal hernias being operated on at the same time or surgery is planned during the follow-up period (incisional and umbilical hernias)
* If hernia recurs within the study period and there is a reoperation within the year
* BMI >40kg/m2
* Patients unable to understand English, written and spoken
* Patients with collagen or connective tissue disorders
* Local (site of surgery) or systemic infection
* Any known diseases that impair nerve function
* Patients who end up getting a mesh repair during surgery
* Impairment of cognitive function (e.g. dementia)
* Pregnancy or lactation
* Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The population under study comprises patients recruited from Shouldice Hospital undergoing inguinal hernia repair. We aim to recruit a sample size of 3,000 patients, males and females, ages 18-90 years, all nationalities and races, capable of speaking and reading English, in good general health, there is no geographic location constraint.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2019-06-17 (Actual); Primary Completion 2023-05-02 (Estimated); Study Completion 2024-05-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with pain severity scores > zero at one year | one-year post surgery
  Brief Pain Inventory - pain severity 0-10 numeric rating scale. Typically score >= 4 corresponds to moderate-to severe pain severity
Proportion of participants with pain-related interference in multiple life domains | one-year post surgery
  Brief Pain Inventory - pain interference
Proportion of participants with neuropathic pain symptoms | one year
  ID Pain 6-items total score ranges from 0 to 6

SECONDARY OUTCOMES:
proportion of participants with significant symptoms of anxiety, depression | one-year post surgery
  Patient Health Questionnaire for Depression and Anxiety - PHQ-4 total score range from 0-12; anxiety subscale 0-6; depression subscale 0-6. total score cutoffs: 0-2 normal; 3-5 mild; 6-8 moderate; 9-12 severe
Do preoperative perceived stress scores predict pain incidence, severity, and/or interference | one-year
  Stress Assessment Test - no norms at present. Scale developed by authors and being validated.
Does pre-operative resilience scores predict lower pain incidence, severity, and/or interference | one-year
  Connor-Davidson Resilience Scale-2. Total score ranges from 0-8. There are no clinical cut-offs for this scale
Do pain preoperative and early postoperative pain catastrophizing scores predict pain incidence, severity, and/or interference | one year
  Pain Catastrophizing Scale -4 item. Total score range: 0-16. There are no sub scales and no cut-offs for this scale

CONTACTS AND LOCATIONS:
Overall Officials: Joel Katz, PhD, Principal Investigator — York University; Robert BenDavid, MD, Principal Investigator — Shouldice Hospital
Locations (1):
- Shouldice Hospital, Thornhill, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mainprize M, Svendrovski A, Paasch C, Yilbas A, Katz J. Matching males and females undergoing Shouldice repair using a prospective, longitudinal design. Can J Surg. 2025 Aug 8;68(4):E325-E332. doi: 10.1503/cjs.012824. Print 2025 Jul-Aug. PMID 40780873